CLINICAL TRIAL: NCT04864509
Title: The Effects of Melatonin Treatment on Bone, Marrow, Sleep and Blood Pressure in Post Menopausal Women
Brief Title: The Effects of Melatonin Treatment on Bone, Marrow, Sleep and Blood Pressure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-AKA
Record Dates: First submitted 2020-08-12; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2020-06

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin 10mg (Active Comparator): Nightly oral dose
  Interventions: Drug: Melatonin 10 MG
- Placebo (Placebo Comparator): nightly oral dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin 10 MG — Nightly dose
  Arms: Melatonin 10mg
Drug: Placebo — Nightly dose
  Arms: Placebo

SUMMARY:
Melatonin protects your bones while losing fat! This was previously demonstrated by our group. The mechanisms behind these findings are still elusive, and the aim of the present study is to assess the mechanisms.

In a double-blinded randomized controlled trial 40 postmenopausal woman are randomized to receive either 10 mg melatonin or placebo nightly for three months. Changes in gene expression in marrow cells will be assessed through micro array. Markers of bone metabolism will be assessed through biochemical markers. Cardiovascular health will be measured by tonometry and 24h blood pressure.

The results of the study will contribute with important knowledge about the beneficial effects of melatonin making it an interesting supplement to known treatment regimens against osteoporosis and overweight.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women between 55 and 75 years

Exclusion Criteria:

* Severely impaired renal function
* Severely impaired hepatic function
* Coagulation factors PP<0.6
* Hypercalcemia (p-ion calcium >1.32 nmol/l)
* Previous or present malignancies (except a treated skin cancer that is not melanoma or treated carcinoma in situ, 2 years since last therapy)
* Diseases affecting the calcium homeostasis including untreated thyroid diseases
* Regular use of medicine affecting the calcium homeostasis, including diuretics, fenemal, lithium, antiepileptica and glucosteroids
* Selective serotonin reuptake inhibitor (SSRI)-products with fluvoxamin
* Treatment with carbamazepin
* Treatment with rifampicin
* Severe malabsorption syndrome including gastric or intestinal resection
* Alcohol or drug abuse
* Smokers

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — self-presentation
Enrollment: 40 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Gene expression | After study completion. Up to one year
  Changes in gene expression in human mesenchymal stem cells.The biopsies are put on freeze after obtaining them. All biopsies are analysed at once.

SECONDARY OUTCOMES:
Biochemical markers | After study completion. Up to one year
  Changes in biochemical markers of bone metabolism measured in blood: Markers include PTH (pmol/l), ionized calcium (mmol/l) CTX (ug/l). Although different units they all contribute to the overall evaluation of bone metabolism and must therefore be regarded as the same outcome measure
Quality of sleep | After study completion. Up to one year
  Assessed through the questionnaire Pittsburgh quality of sleep questionnaire. A validated questionnaire assessing the quality of sleep. A score between 0-5 indicates a good quality of sleep. Scores above 5 indicate a poor quality of sleep.
Cardiovascular health | After study completion. Up to one year
  Changes in 24h blood pressure and arterial stiffness measured by standardized equipment

CONTACTS AND LOCATIONS:
Overall Officials: Anne Kristine Amstrup, Principal Investigator — Aarhus University Hospital